CLINICAL TRIAL: NCT03419962
Title: Changes in Health and Functional Status in Patients With Chronic Obstructive Pulmonary Disease (COPD) During Therapy With Spiolto® Respimat® [ELLACTO]
Brief Title: Greek NIS Spiolto ELLACTO
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0073
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COPD patients: Chronic obstructive pulmonary disease
  Interventions: Drug: MaxSpiolto® Respimat® 160 Characters...

INTERVENTIONS:
Drug: MaxSpiolto® Respimat® 160 Characters... — as per the approved SmPC
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO

SUMMARY:
Open-label observational study: including COPD patients receiving treatment with Spiolto® Respimat® for approximately 6 weeks, which is the average time between two medical consultations

ELIGIBILITY:
Inclusion Criteria:

* Therapeutic indication before entering the enrollment face is patients diagnosed with COPD requiring a combination therapy of two long-acting bronchodilators (LAMA + LABA) according to approved SmPC and guidelines, COPD GOLD 2017 groups B to D
* Female and male patients ≥40 years of age
* Treatment with Spiolto ® Respimat® acc. to SmPC and at the discretion of the physician
* Written informed consent prior to participation

Exclusion Criteria:

* Patients with contraindications according to Spiolto® Respimat® SmPC
* Patients who have been treated with a LABA/LAMA combination (free and fixed dose) in the previous 6 weeks or patients already on a combination of LAMA and LABA therapy; either as a fixed combination product or as separate components Note: Patients previously treated with LABA or LAMA (with or without ICS) are eligible to be included in the study
* Patients continuing LABA-ICS treatment should not be additionally treated with Spiolto® Respimat® in order to avoid a double dosing of long-acting beta-agonists
* Patients for whom further follow-up is not possible at the enrolling site during the planned study period of approx. 6 weeks
* Pregnancy and lactation
* Patients currently listed for lung transplantation
* Current participation in any clinical trial or any other non-interventional study of a drug or device

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1300 patients with chronic obstructive pulmonary disease (COPD) in whom combination treatment with long-acting bronchodilators is indicated in accordance with the guidelines are to be observed by approx. 100 pulmonologists in the setting of private practice. The NIS will take place in Greece and sites in urban as well as rural areas will be included. The nationwide distribution of the participating pulmonologists as well as the number of patients enrolled are intended to ensure that the data collected are representative.
Sampling Method: Probability Sample
Enrollment: 1360 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Greece (15):
  - Metropolitan, Aegina
  - Metroplitan, Athens
  - Metropolitan, Athens
  - Metropolitan, Chania
  - Metropolitan, Heraklio
  - Metropolitan, Hrakleio
  - Metropolitan, Hraklio
  - Diavalkaniko, Ioannina
  - Diavalkaniko, Kavala
  - Diavalkaniko, Larissa
  - Metropolitan, Pátrai
  - Diavalkaniko, Serres
  - Merkouropoulos Markos, Thessaloniki
  - Diavalkaniko, Thessaloniki
  - Diavalkaniko, Volos

REFERENCES:
- [Derived] Kosmas E, Titopoulos I, Patentalakis G, Nikas N. An Observational Study Assessing Changes in Health and Functional Status in Patients with Chronic Obstructive Pulmonary Disease (COPD) During Therapy with Spiolto(R) Respimat(R) in Everyday Clinical Practice: The Greek ELLACTO Study. Pulm Ther. 2021 Dec;7(2):429-443. doi: 10.1007/s41030-021-00156-7. Epub 2021 May 3. PMID 33939158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label observational study to measure the effectiveness of 6 weeks treatment of Spiolto® Respimat® in Patients with Chronic Obstructive Pulmonary Disease (COPD). The Clinical COPD Questionnaire (CCQ)-score was used to evaluate changes in health and functional status.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that all participants met all inclusion and non of the exclusion criteria. 1 enrolled participant was excluded as he/she did not have at least one documented administration of Spiolto® Respimat®.
Groups:
- Spiolto® Respimat® 2.5mg/2.5mg: 2.5microgram/2.5 microgram of Spiolto® Respimat® (tiotropium/olodaterol) was orally administered once daily via the Respimat inhaler over 6 weeks in patients with chronic obstructive pulmonary disease (COPD).
Period: Overall Study
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
Started | 1359
Completed | 1322
Not Completed | 37
Not completed — Change to other medication | 1
Not completed — Refusal of continuing with trial drug | 1
Not completed — Lost to Follow-up | 3
Not completed — Difficulty in inhaling the doses | 1
Not completed — Missing completion data | 31

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): Treated set included all screened patients with the informed consent, date of registration and at least one documented administration of Spiolto® Respimat®.
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
Number analyzed (Participants) | 1359
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Set (TS): Treated Set included all screened patients with the informed consent, date of registration and at least one documented administration of Spiolto® Respimat®.
  Years | 68.1 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set: Treated Set included all screened patients with the informed consent, date of registration and at least one documented administration of Spiolto® Respimat®.
  Participants
    Female | 437
    Male | 922
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving "Therapeutic Success" Defined as a ≥ 0.4 Point of Decrease in the Clinical COPD Questionnaire (CCQ) Score
Description: Therapeutic success was defined as ≥0.4 point decrease in the Clinical COPD Questionnaire (CCQ) score between visit 1 (baseline visit at study start) and visit 2 (final visit at end of study, approximately 6 weeks after visit 1).
  The CCQ contained 10 questions about symptoms, functional status and mental status. Each of the 10 CCQ questions was scored by the patient on a 7-point scale (ranging between 0=asymptomatic/no-limitation, to 6=symptomatic/totally limited). The sum of the scores divided by 10 gives the CCQ score. A higher CCQ score is indicative of worse status. A decrease of 0.4 points is considered to be the minimal clinically important difference (MCID) for CCQ score.
Time Frame: Between visit 1 (baseline visit at study start) and visit 2 (final visit after end of study, approximately 6 weeks after visit 1).
Population: Full Analysis Set (FAS): The FAS comprised all patients of the Treated Set (TS) with a completed CCQ score at both visit 1 and visit 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
Number analyzed (Participants) | 1332
Percentage of participants | 64.3 [62 to 67]

2. Secondary Outcome: Absolute Change in Clinical COPD Questionnaire (CCQ) Score Between Visit 1 and Visit 2
Description: Absolute change in Clinical COPD Questionaire (QQC) score between visit 1 (baseline visit at study start) and visit 2 (final visit at end of study, approximately 6 weeks after visit 1).
  The CCQ contained 10 questions about symptoms, functional status and mental status. Each of the 10 CCQ questions was scored by the patient on a 7-point scale between 0 and 6. The sum of the scores divided by 10 gives the CCQ score which measured the health and functional status. A higher CCQ score is indicative of worse status.
Time Frame: At visit 1 (baseline visit at study start) and at visit 2 (final visit at end of study, approximately 6 weeks after visit 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CCQ-score
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
Number analyzed (Participants) | 1332
CCQ-score | -0.63 (0.635)

3. Secondary Outcome: Absolute Change in the Functional Status Subdomain of Clinical COPD Questionnaire (CCQ-4) Score Between Visit 1 and Visit 2
Description: Absolute change in the functional status subdomain of Clinical COPD Questionnaire (CCQ-4) score between visit 1 (baseline visit at study start) and visit 2 (final visit at end of study, approximately 6 weeks after visit 1).
  The CCQ-4 score is a subdomain of the CCQ-score. It contains 4 questions about the functional status of patients. Each questions was scored by the patient on a 7-point scale, (ranging between 0=asymptomatic/no-limitation, to 6=symptomatic/totally limited). The QQC-4 score was calculated by the sum of 4 questions divided by 4. A higher CCQ-4 score was indicative of worse status.
Time Frame: At visit 1 (baseline visit at study start) and at visit 2 (final visit at the end of study, approximately 6 weeks after visit 1).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CCQ-4 score
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
Number analyzed (Participants) | 1332
CCQ-4 score | -0.59 (0.714)

4. Secondary Outcome: General Condition of Patient at Visit 1 and Visit 2
Description: General condition of the patient, evaluated by Physician´s Global Evaluation (PGE) score at visit 1 and visit 2.
  The PGE score uses a eight-point ordinal scale, ranging from poor (1,2) to excellent (7,8).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
Number analyzed (Participants) | 1332
Participants
  Visit 1: Poor (1-2) | 153
  Visit 1: Satisfactory (3-4) | 496
  Visit 1: Good (5-6) | 568
  Visit 1: Excellent (7-8) | 115
  Visit 1: Missing (Not Done) | 0
  Visit 2: Poor (1-2) | 38
  Visit 2: Satisfactory (3-4) | 260
  Visit 2: Good (5-6) | 709
  Visit 2: Excellent (7-8) | 323
  Visit 2: Missing (Not Done) | 2

5. Secondary Outcome: Patients Satisfaction With Spiolto® Respimat® at Visit 2
Description: The patients satisfaction with Respimat was assessed at end of study (visit 2) by the Patient Satisfaction and Preference Questionnaire (PASAPQ) Part 1. PASAPQ Part 1 uses a 7-point ordinal scale, ranging from very dissatisfied to very satisfied, to rate the satisfaction with inhaler attributes. The patients were requested to describe their satisfaction level answering three questions.
Time Frame: At visit 2 (final visit, at the end of study, approximately 6 weeks after baseline visit).
Population: Full Analysis Set (FAS): The FAS comprised all patients of the Treated Set (TS) with a completed CCQ score at both visit 1 and visit 2. Only 1330 patients completed the PASAPQ Part1+Part2.
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
Number analyzed (Participants) | 1332
Participants
  Satisfaction with feeling of inhaled dose: Very dissatisfied | 2
  Satisfaction with feeling of inhaled dose: Dissatisfied | 7
  Satisfaction with feeling of inhaled dose: Somewhat dissatisfied | 7
  Satisfaction with feeling of inhaled dose: Neither satisfied nor dissatisfied | 99
  Satisfaction with feeling of inhaled dose: Somewhat satisfied | 184
  Satisfaction with feeling of inhaled dose: Satisfied | 600
  Satisfaction with feeling of inhaled dose: Very satisfied | 432
  Satisfaction with feeling of inhaled dose: Missing | 1
  Satisfaction with reliability of inhaler: Very dissatisfied | 4
  Satisfaction with reliability of inhaler: Dissatisfied | 0
  Satisfaction with reliability of inhaler: Somewhat dissatisfied | 13
  Satisfaction with reliability of inhaler: Neither satisfied nor dissatisfied | 71
  Satisfaction with reliability of inhaler: Somewhat satisfied | 190
  Satisfaction with reliability of inhaler: Satisfied | 647
  Satisfaction with reliability of inhaler: Very satisfied | 406
  Satisfaction with reliability of inhaler: Missing | 1
  Satisfaction with ease of inhaling: Very dissatisfied | 3
  Satisfaction with ease of inhaling: Dissatisfied | 6
  Satisfaction with ease of inhaling: Somewhat dissatisfied | 8
  Satisfaction with ease of inhaling: Neither satisfied nor dissatisfied | 67
  Satisfaction with ease of inhaling: Somewhat satisfied | 175
  Satisfaction with ease of inhaling: Satisfied | 614
  Satisfaction with ease of inhaling: Very satisfied | 458
  Satisfaction with ease of inhaling: Missing | 1

6. Secondary Outcome: Patients Preference for Spiolto® Respimat® at Visit 2
Description: Patients preference for Respimat® Inhaler vs. Spiriva HandiHaler (HH) was assessed using the abbreviated Patient Satisfaction and Preference Questionnaire (PASAPQ) Part 2 survey. Patients were requested to describe their preference for each inhaler device by answering 2 additional questions.
Time Frame: At visit 2 (final visit, at the end of study, approximately 6 weeks after baseline visit)
Population: Only patients from the Full Analysis Set (FAS), who have used Spiriva HandiHaler (HH) prior to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
Number analyzed (Participants) | 254
Participants
  Preference for Spiriva HH | 17
  Preference for Spiolto Respimat | 217
  No preference | 20

7. Secondary Outcome: Patient's Willingness to Continue Treatment With Spiolto® Respimat® at Visit 2
Description: Patients' reported willingness to continue using either of the inhalers was measured with a scale score ranking from 0 to 100. 0 indicates not willing to continue using this inhaler and 100 indicates definitely willing to continue using it.
Time Frame: At visit 2 (final visit, at the end of study, approximately 6 weeks after baseline visit).
Population: Only patients from the Full Analysis Set (FAS), who have used Spiriva HandiHaler (HH) prior to the study. Only 253 patients were analyzed, as one patient did not answer the question.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
Number analyzed (Participants) | 253
Scores on scale
  Scoring of Spiriva HH | 32.3 (27.06)
  Scoring of Spiolto® Respimat® | 79.8 (21.19)

ADVERSE EVENTS:
Time Frame: From study start until end of study, up to 6 weeks.
Description: Adverse Events were reported for the Treated Set (TS). TS included all screened patients with the informed consent, date of registration and at least one documented administration of Spiolto® Respimat®.
Arm/Group | Spiolto® Respimat® 2.5mg/2.5mg
All-Cause Mortality (participants affected / at risk) | 0/1359
Serious Adverse Events (participants affected / at risk) | 1/1359
Other Adverse Events (participants affected / at risk) | 0/1359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiolto® Respimat® 2.5mg/2.5mg (N=1359)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT03419962/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT03419962/SAP_001.pdf